CLINICAL TRIAL: NCT00661674
Title: Examination of Palonosetron and Hydroxyzine Pre-treatment as a Possible Method to Reduce the Objective Signs of Experimentally-induced Acute Opioid Withdrawal in Humans: a Double-blind, Randomized, Placebo-controlled Crossover Study
Brief Title: Palonosetron and Hydroxyzine to Reduce Opioid Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Larry Fu-nien Chu, Professor of Anesthesia, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-04152008-1099
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Substance-Related Disorders
Keywords: Palonosetron; Hydroxyzine; Acute opioid withdrawal
MeSH Terms: conditions — Substance-Related Disorders | interventions — Palonosetron; Hydroxyzine

STUDY DESIGN:
Intervention Model Description: There were three treatment arms to the study: Placebo, Palonosetron, and Palonosetron + Hydroxyzine (Combo). Participants were not randomized in between these arms, all participants completed each arm of the study in a cross-over study methodology (Placebo, Palonosetron, Palonosetron + Hydroxyzene (combo). Participants were individually randomized into the order in which they participated in each arm.
  Per sequence each individual participant underwent the following randomization schedule:
  Participant 1: Placebo, Combo, Palonosetron Participant 2: Palonosetron, Combo, Placebo Participant 3: Palonosetron, Combo, Placebo Participant 4: Combo, Placebo, Palonosetron Participant 5: Placebo, Palonosetron, Combo Participant 6: Combo, Palonosetron, Placebo Participant 7: Combo, Placebo, Palonosetron Participant 8: Combo, Palonosetron, Placebo Participant 9: Palonosetron, Placebo, Combo Participant 10: Placebo, Combo, Palonosetron
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1: Placebo, Combo, Palonosetron (Experimental): At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Placebo
  Week 2: Palonosetron + Hydroxyzine Combo
  Week 3: Palonosetron
  Interventions: Drug: Palonosetron; Drug: Hydroxyzine; Other: Placebo
- Sequence 2: Palonosetron, Combo, Placebo (Experimental): At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Palonosetron
  Week 2: Palonosetron + Hydroxyzine Combo
  Week 3: Placebo
  Interventions: Drug: Palonosetron; Drug: Hydroxyzine; Other: Placebo
- Sequence 3: Combo, Placebo, Palonosetron (Experimental): At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Palonosetron + Hydroxyzine Combo
  Week 2: Placebo
  Week 3: Palonosetron
  Interventions: Drug: Palonosetron; Drug: Hydroxyzine; Other: Placebo
- Sequence 4: Placebo, Palonosetron, Combo (Experimental): At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Placebo
  Week 2: Palonosetron only
  Week 3: Palonosetron + Hydroxyzine Combo
  Interventions: Drug: Palonosetron; Drug: Hydroxyzine; Other: Placebo
- Sequence 5: Combo, Palonosetron, Placebo (Experimental): At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Palonosetron + Hydroxyzine Combo
  Week 2: Palonosetron only
  Week 3: Placebo
  Interventions: Drug: Palonosetron; Drug: Hydroxyzine; Other: Placebo
- Sequence 6: Palonosetron, Placebo, Combo (Experimental): At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Palonosetron only
  Week 2: Placebo
  Week 3:Palonosetron + Hydroxyzine Combo
  Interventions: Drug: Palonosetron; Drug: Hydroxyzine; Other: Placebo

INTERVENTIONS:
Drug: Palonosetron — Over 3 study visits, patients will receive one of the following treatment regimens:
  * Placebo saline IV and sugar pill
  * 0.75 mg Palonosetron IV and sugar pill
  * 0.75 mg Palonosetron IV and 100 mg hydroxyzine PO
  Other Names: Aloxi
Drug: Hydroxyzine — Over 3 study visits, patients will receive one of the following treatment regimens:
  * Placebo saline IV and sugar pill
  * 0.75 mg Palonosetron IV and sugar pill
  * 0.75 mg Palonosetron IV and 100 mg hydroxyzine PO
  Other Names: Vistaril, Atarax
Other: Placebo — Over 3 study visits, patients will receive one of the following treatment regimens:
  * Placebo saline IV and sugar pill
  * 0.75 mg Palonosetron IV and sugar pill
  * 0.75 mg Palonosetron IV and 100 mg hydroxyzine PO

SUMMARY:
Opioid medications are commonly used for pain relief. When given over time, physical dependence can occur. This results in unpleasant side effects--such as agitation and nausea--if opioid medications are suddenly stopped. We are interested in knowing if a medication named Ondansetron can help ease or prevent symptoms associated with opioid withdrawal. We are also interested in knowing if a similar (but more potent FDA-approved drug, palonosetron) can more effectively treat withdrawal symptoms with or without combination with an antihistamine called hydroxyzine (vistaril).

DETAILED DESCRIPTION:
We hope to learn if Palonosetron and/or combination with hydroxyzine can be used to prevent or attenuate the signs and symptoms of opioid withdrawal. If we find that it can help prevent these symptoms, it may become a new treatment that can aid patients suffering from these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Ages 18-35
* No allergies to morphine or palonosetron
* No history of addiction or substance abuse

Exclusion Criteria:

* Female
* Younger than 18 or older than 35
* History of substance abuse
* Raynaud's disease or coronary artery disease
* Allergies to morphine or palonosetron

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Larry Fu-nien Chu, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Advancing Pain Research Care and Education, Board on Health Sciences Policy, Institute of Medicine. A call for cultural transformation of attitudes toward pain and its prevention and management. J Pain Palliat Care Pharmacother. 2011;25(4):365-9. doi: 10.3109/15360288.2011.621516. PMID 22126167
- [Background] Kuehn BM. Opioid prescriptions soar: increase in legitimate use as well as abuse. JAMA. 2007 Jan 17;297(3):249-51. doi: 10.1001/jama.297.3.249. No abstract available. PMID 17227967
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Kobinger W, Walland A. Investigations into the mechanism of the hypotensive effect of 2-(2,6-dichlorphenylamino)-2-imidazoline-HCl. Eur J Pharmacol. 1967 Dec;2(3):155-62. doi: 10.1016/0014-2999(67)90080-5. No abstract available. PMID 5626889
- [Background] Chu LF, Liang DY, Li X, Sahbaie P, D'arcy N, Liao G, Peltz G, David Clark J. From mouse to man: the 5-HT3 receptor modulates physical dependence on opioid narcotics. Pharmacogenet Genomics. 2009 Mar;19(3):193-205. doi: 10.1097/FPC.0b013e328322e73d. PMID 19214139
- [Background] Costall B, Jones BJ, Kelly ME, Naylor RJ, Onaivi ES, Tyers MB. Sites of action of ondansetron to inhibit withdrawal from drugs of abuse. Pharmacol Biochem Behav. 1990 May;36(1):97-104. doi: 10.1016/0091-3057(90)90132-2. PMID 2140900
- [Background] Gulati A, Bhargava HN. Brain and spinal cord 5-HT2 receptors of morphine-tolerant-dependent and -abstinent rats. Eur J Pharmacol. 1989 Aug 22;167(2):185-92. doi: 10.1016/0014-2999(89)90578-5. PMID 2591474
- [Background] Tao R, Ma Z, Auerbach SB. Alteration in regulation of serotonin release in rat dorsal raphe nucleus after prolonged exposure to morphine. J Pharmacol Exp Ther. 1998 Jul;286(1):481-8. PMID 9655893
- [Background] Ingram SL, Vaughan CW, Bagley EE, Connor M, Christie MJ. Enhanced opioid efficacy in opioid dependence is caused by an altered signal transduction pathway. J Neurosci. 1998 Dec 15;18(24):10269-76. doi: 10.1523/JNEUROSCI.18-24-10269.1998. PMID 9852564
- [Background] Tao R, Auerbach SB. Involvement of the dorsal raphe but not median raphe nucleus in morphine-induced increases in serotonin release in the rat forebrain. Neuroscience. 1995 Sep;68(2):553-61. doi: 10.1016/0306-4522(95)00154-b. PMID 7477965
- [Background] Pinelli A, Trivulzio S, Tomasoni L. Effects of ondansetron administration on opioid withdrawal syndrome observed in rats. Eur J Pharmacol. 1997 Dec 11;340(2-3):111-9. doi: 10.1016/s0014-2999(97)01349-6. PMID 9537805
- [Background] Smith HS, Cox LR, Smith EJ. 5-HT3 receptor antagonists for the treatment of nausea/vomiting. Ann Palliat Med. 2012 Jul;1(2):115-20. doi: 10.3978/j.issn.2224-5820.2012.07.07. PMID 25841471
- [Background] Compton P, Miotto K, Elashoff D. Precipitated opioid withdrawal across acute physical dependence induction methods. Pharmacol Biochem Behav. 2004 Feb;77(2):263-8. doi: 10.1016/j.pbb.2003.10.017. PMID 14751453
- [Background] Grunberg SM, Koeller JM. Palonosetron: a unique 5-HT3-receptor antagonist for the prevention of chemotherapy-induced emesis. Expert Opin Pharmacother. 2003 Dec;4(12):2297-303. doi: 10.1517/14656566.4.12.2297. PMID 14640928
- [Background] Mustian KM, Devine K, Ryan JL, Janelsins MC, Sprod LK, Peppone LJ, Candelario GD, Mohile SG, Morrow GR. Treatment of Nausea and Vomiting During Chemotherapy. US Oncol Hematol. 2011;7(2):91-97. doi: 10.17925/ohr.2011.07.2.91. PMID 24466408
- [Background] Smith HS, Laufer A. Opioid induced nausea and vomiting. Eur J Pharmacol. 2014 Jan 5;722:67-78. doi: 10.1016/j.ejphar.2013.09.074. Epub 2013 Oct 21. PMID 24157979
- [Background] Mazurkiewicz-Kwilecki IM, Bielkiewicz B. The effects of chronic morphine treatment on histamine concentration and histidine decarboxylase activity in rat brain. Prog Neuropsychopharmacol. 1978;2(1):93-9. doi: 10.1016/0364-7722(78)90027-9. No abstract available. PMID 569343
- [Background] Wong CL, Roberts MB. The possible role of brain histamine and H1 and H2 receptors in the development of morphine tolerance and physical dependence in mice. Agents Actions. 1975 Dec;5(5):476-83. doi: 10.1007/BF01972684. PMID 1241224
- [Background] Wong CL, Roberts MB. The effects of L-histidine and of specific histamine receptor agonists, on the expression of morphine tolerance and physical dependence in mice. Agents Actions. 1976 Sep;6(5):569-76. doi: 10.1007/BF01971571. PMID 987696
- [Background] Hoehe M. Influence of the menstrual cycle on neuroendocrine and behavioral responses to an opiate agonist in humans: preliminary results. Psychoneuroendocrinology. 1988;13(4):339-44. doi: 10.1016/0306-4530(88)90059-5. PMID 2852375
- [Background] Handelsman L, Cochrane KJ, Aronson MJ, Ness R, Rubinstein KJ, Kanof PD. Two new rating scales for opiate withdrawal. Am J Drug Alcohol Abuse. 1987;13(3):293-308. doi: 10.3109/00952998709001515. PMID 3687892
- [Background] Alsaadi SM, McAuley JH, Hush JM, Lo S, Lin CW, Williams CM, Maher CG. Poor sleep quality is strongly associated with subsequent pain intensity in patients with acute low back pain. Arthritis Rheumatol. 2014 May;66(5):1388-94. doi: 10.1002/art.38329. PMID 24782195
- [Background] Schuh-Hofer S, Wodarski R, Pfau DB, Caspani O, Magerl W, Kennedy JD, Treede RD. One night of total sleep deprivation promotes a state of generalized hyperalgesia: a surrogate pain model to study the relationship of insomnia and pain. Pain. 2013 Sep;154(9):1613-1621. doi: 10.1016/j.pain.2013.04.046. Epub 2013 May 11. PMID 23707287
- [Background] De Leon A. Palonosetron (Aloxi): a second-generation 5-HT(3) receptor antagonist for chemotherapy-induced nausea and vomiting. Proc (Bayl Univ Med Cent). 2006 Oct;19(4):413-6. doi: 10.1080/08998280.2006.11928210. PMID 17106506
- [Background] Boon JH, Hopkins D. Hydroxyzine premedication--does it provide better anxiolysis than a placebo? S Afr Med J. 1996 Jun;86(6):661-4. PMID 8764421
- [Background] Roychoudhury M, Kulkarni SK. Prevention of morphine discontinuation phenomenon in mice by ondansetron, a selective 5-HT3 antagonist. Methods Find Exp Clin Pharmacol. 1996 Dec;18(10):677-83. PMID 9121224
- [Background] Cui R, Suemaru K, Li B, Kohnomi S, Araki H. Tropisetron attenuates naloxone-induced place aversion in single-dose morphine-treated rats: role of alpha7 nicotinic receptors. Eur J Pharmacol. 2009 May 1;609(1-3):74-7. doi: 10.1016/j.ejphar.2008.12.051. Epub 2009 Jan 17. PMID 19374878
- [Background] Araki H, Kawakami KY, Jin C, Suemaru K, Kitamura Y, Nagata M, Futagami K, Shibata K, Kawasaki H, Gomita Y. Nicotine attenuates place aversion induced by naloxone in single-dose, morphine-treated rats. Psychopharmacology (Berl). 2004 Feb;171(4):398-404. doi: 10.1007/s00213-003-1595-7. Epub 2003 Sep 10. PMID 13680070
- [Background] Motoshima S, Suemaru K, Kawasaki Y, Jin C, Kawasaki H, Gomita Y, Araki H. Effects of alpha4beta2 and alpha7 nicotinic acetylcholine receptor antagonists on place aversion induced by naloxone in single-dose morphine-treated rats. Eur J Pharmacol. 2005 Sep 5;519(1-2):91-5. doi: 10.1016/j.ejphar.2005.06.050. PMID 16098507
- [Background] Maricq AV, Peterson AS, Brake AJ, Myers RM, Julius D. Primary structure and functional expression of the 5HT3 receptor, a serotonin-gated ion channel. Science. 1991 Oct 18;254(5030):432-7. doi: 10.1126/science.1718042.
- [Background] Albertson TE, Chenoweth J, Ford J, Owen K, Sutter ME. Is it prime time for alpha2-adrenocepter agonists in the treatment of withdrawal syndromes? J Med Toxicol. 2014 Dec;10(4):369-81. doi: 10.1007/s13181-014-0430-3. PMID 25238670
- [Background] Walsh SL, Strain EC, Bigelow GE. Evaluation of the effects of lofexidine and clonidine on naloxone-precipitated withdrawal in opioid-dependent humans. Addiction. 2003 Apr;98(4):427-39. doi: 10.1046/j.1360-0443.2003.00372.x. PMID 12653813
- [Derived] Erlendson MJ, D'Arcy N, Encisco EM, Yu JJ, Rincon-Cruz L, Peltz G, Clark JD, Chu LF. Palonosetron and hydroxyzine pre-treatment reduces the objective signs of experimentally-induced acute opioid withdrawal in humans: a double-blinded, randomized, placebo-controlled crossover study. Am J Drug Alcohol Abuse. 2017 Jan;43(1):78-86. doi: 10.1080/00952990.2016.1210614. Epub 2016 Aug 11. PMID 27712113

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Placebo, Combo, Palonosetron: At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Placebo
  Week 2: Combo
  Week 3: Palonosetron
- Sequence 2: Palonosetron, Combo, Placebo: At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Palonosetron
  Week 2: Combo
  Week 3: Placebo
- Sequence 3: Combo, Placebo, Palonosetron: At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Combo
  Week 2: Placebo
  Week 3: Palonosetron
- Sequence 4: Placebo, Palonosetron, Combo: At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Placebo
  Week 2: Palonosetron
  Week 3: Combo
- Sequence 5: Combo, Palonosetron, Placebo: At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Combo
  Week 2: Palonosetron
  Week 3: Placebo
- Sequence 6: Palonosetron, Placebo, Combo: At T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with either placebo (0.9% normal saline), palonosetron IV (0.75mg), or palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
  Week 1: Palonosetron
  Week 2: Placebo
  Week 3: Combo
Period: Overall Study
Arm/Group | Sequence 1: Placebo, Combo, Palonosetron | Sequence 2: Palonosetron, Combo, Placebo | Sequence 3: Combo, Placebo, Palonosetron | Sequence 4: Placebo, Palonosetron, Combo | Sequence 5: Combo, Palonosetron, Placebo | Sequence 6: Palonosetron, Placebo, Combo
Started (Only 1 intervention per sequence was given each week based on sequence assignment) | 2 (Participants 1 & 10 were assigned to sequence 1) | 2 (Participants 2 & 3 were assigned to sequence 2) | 2 (Participants 4 & 7 were assigned to sequence 3) | 1 (Participant 5 was assigned to sequence 4) | 2 (Participants 6 & 8 were assigned to sequence 5) | 1 (Participant 9 was assigned to sequence 6)
Completed | 2 (Participants 1 & 10 completed sequence 1) | 2 (Participants 2 & 3 completed sequence 2) | 2 (Participants 4 & 7 completed sequence 3) | 1 (Participant 5 completed sequence 4) | 2 (Participants 6 & 8 completed sequence 5) | 1 (Participant 9 completed sequence 6)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 10 healthy male volunteers recruited from the San Francisco Bay Area. All study sessions took place at the Stanford University School of Medicine, Department of Anesthesia.
Groups:
- Overall Study: Over three study sessions each spaced one week apart participants received either placebo IV + PO, Palonosetron IV (0.75 mg) + placebo PO, or Palonosetron IV (0.75 mg) + Hydroxyzine PO (100mg).
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (2.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: OOWS Score
Description: The OOWS is a 13-item instrument documenting physically observable signs of withdrawal, which are rated as present (1) or absent (0) during the observation period. Maximum score possible = 13, minimum score possible = 0. T=15 minutes post naloxone administration coordinates with T = 180 (min) for the entire study session.
  OOWS scores at T=180 is the primary outcome measure of the study compared with baseline OOWS scores at T=-30 (30 minutes prior to study medication administration). Reported time frames are in relation to time past since administration of study medications.
  Mean post-Naloxone OOWS scores (+/- SEM) were determined for pretreatment groups
Time Frame: Change from baseline in OOWS score at 180 minutes (15 minutes post naloxone administration)
Measure: Mean (Standard Error); unit: units on a scale (OOWS Scale)
Groups:
- Placebo: Each participant had one session in which they received a placebo tablet pretreatment prior to naloxone-precipitated withdrawal.
- Palonosetron: Each participant had one session in which they received palonosetron IV pretreatment prior to naloxone-precipitated withdrawal.
- Palonosetron + Hydroxyzine: Each participant had one session in which they received IV palonosetron + PO hydroxyzine pretreatment prior to naloxone-precipitated withdrawal.
Arm/Group | Placebo | Palonosetron | Palonosetron + Hydroxyzine
Number analyzed (Participants) | 10 | 10 | 10
units on a scale (OOWS Scale) | 3.5 (0.76) | 1.0 (0.37) | 0 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Palonosetron vs Palonosetron + Hydroxyzine; Null Hypothesis: There will be no difference in OOWS scores when comparing treatment groups (Palonosetron & Palonosetron + Hydroxyzine) with placebo. Analysis of the data obtained in our prior study indicated that analysis of 10 individuals would provide 90% power to detect a treatment effect. Therefore, we examined the effect of three different pretreatments on naloxone-induced opiate withdrawal signs in 10 healthy individuals; Test type: Superiority or Other; p = 0.0001, Friedman Test — p-value represents comparison between OOWS scores at T=180 and the baseline measurements at T=-30

2. Secondary Outcome: SOWS Score
Description: The SOWS score is composed of 16 subjective symptoms rated on a scale of 0 to 4 (0=not at all, 4=extremely) based on what subjects were experiencing at the time of testing. 15 minutes post naloxone administration coordinates with T = 180 (min) for the entire study session.
  The highest score possible (64) would indicate that the individual was experiencing every symptom of opioid withdrawal to the fullest extent possible while the lowest score (0) would indicate that the individual was not experiencing any symptoms of opioid withdrawal.
  Mean post-naloxone SOWS scores (+/- SEM) were computed for pretreatment groups: Placebo, palonosetron, and palonosetron with hydroxyzine
Time Frame: Change from baseline in SOWS score at 180 minutes (15 minutes post naloxone administration)
Measure: Mean (Standard Error); unit: units on a scale (SOWS Scale)
Arm/Group | Placebo | Palonosetron | Palonosetron + Hydroxyzine
Number analyzed (Participants) | 10 | 10 | 10
units on a scale (SOWS Scale) | 6.0 (1.86) | 4.0 (1.86) | 3.5 (1.39)
Statistical Analysis 1: Comparison: Placebo vs Palonosetron vs Palonosetron + Hydroxyzine; Null Hypothesis: There will be no difference in SOWS scores when comparing the 2 treatment groups (Palonosetron & Palonosetron + Hydroxyzine) with placebo. Analysis of the data obtained in our prior study indicated that analysis of 10 individuals would provide 90% power to detect a treatment effect. Therefore, we examined the effect of three different pretreatments on naloxone-induced opiate withdrawal signs in 10 healthy individuals; Test type: Superiority or Other; p = 0.2244, Friedman Test — p-value represents comparison between SOWS scores at T=180 and the baseline measurements at T=-30

ADVERSE EVENTS:
Time Frame: Data on adverse events was recorded throughout the duration of the study including study session #1 (week 1), study session #2 (week 2) and study session #3 (week 3).
Groups:
- Placebo: At timepoint T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with placebo (0.9% normal saline) in a crossover study design. Participants returned for three study sessions, each one week apart to receive all three study combinations. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
- Palonosetron + Placebo: At timepoint T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with palonosetron IV (0.75mg) in a crossover study design. Participants returned for three study sessions, each one week apart to receive all three study drug combinations. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
- Palonosetron + Hydroxyzine: At timepoint T = 0 (minutes), healthy (non-opioid dependent, non-substance abuser) male volunteers (N=10) were pre-treated with palonosetron IV (0.75mg) and hydroxyzine per os (PO) (100mg) in a crossover study design. Participants returned for three study sessions, each one week apart to receive all three study combinations. This was followed at T = 30 by intravenous morphine (10mg/70kg). At T = 165, 10mg/70kg naloxone IV was given to precipitate opioid withdrawal. The objective opioid withdrawal score (OOWS) and subjective opioid withdrawal score (SOWS) were determined 5 and 15 minutes after naloxone administration (T = 170, 180, respectively). Baseline measurements were recorded at T = -30 and T = -15.
Arm/Group | Placebo | Palonosetron + Placebo | Palonosetron + Hydroxyzine
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Results are not necessarily generalizable to patients with chronic opioid exposure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No